CLINICAL TRIAL: NCT04775108
Title: First-In-Human Clinical Study for Treatment of Severe Mitral Valve INsufficiency With Epygon™ TRanscatheter Mitral VAlve System (MINERVA FIH)
Brief Title: First-In-Human Clinical Study for Treatment of Severe Mitral Valve INsufficiency With Epygon™ TRanscatheter Mitral VAlve System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Epygon (Industry)
Responsible Party: Sponsor
Organization: Affluent Medical (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MINERVA FIH
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Mitral Valve Regurgitation
Keywords: Mitral regurgitation; Mitral valve replacement
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implanted patients (Experimental): Implantation of Epygon mitral valve prosthesis
  Interventions: Device: Epygon™ Transcatheter Mitral Valve System

INTERVENTIONS:
Device: Epygon™ Transcatheter Mitral Valve System — The EPYGON VALVE is an innovative mitral valve, intended for valve replacement of a native mitral valve through a minimally invasive implant procedure by means of a dedicated implant device.
  The EPYGON VALVE is a bio prosthesis, composed by a functional assembly of bovine pericardium on a NiTinol stent.

SUMMARY:
The EPYGON VALVE is an innovative mitral valve, intended for valve replacement of a native mitral valve through a minimally invasive implant procedure by means of a dedicated implant device.

The EPYGON VALVE is a bio prosthesis, composed by a functional assembly of bovine pericardium on a NiTinol stent.

The purpose of this trial is to assess the safety and feasibility of the Epygon™ Transcatheter mitral valve and the transapical delivery system, in adult patients with severe, symptomatic mitral regurgitation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of age ≥ 60 years.
2. Patients with primary or secondary severe symptomatic mitral valve regurgitation.
3. Patients with severe, symptomatic mitral regurgitation and who have been evaluated by a multidisciplinary Heart Team and deemed to be ineligible for conventional valve surgery and not eligible for transcatheter repair.
4. Patients with a left ventricular ejection fraction ≥ 30%.
5. Patients in NYHA functional classes III to IV.
6. Patients who have clearly accepted participation in this clinical study and who have signed the informed consent.
7. Patients who are willing to accept and undergo all protocol related requirements.
8. Patients not planning to transfer abroad.

Exclusion Criteria:

- Clinical exclusion criteria (preoperative screening)

1. Patients involved in other clinical assessments for drugs or devices that could interfere or alter the study endpoints.
2. Patients with clinical/anatomical conditions unsuitable for a transapical surgical approach.
3. Patients who have previously undergone implantation of a transcatheter aortic valve prosthesis.
4. Patients with previous implantation of a mitral heart valve prosthesis.
5. Patients with previous implantation of a mitral annuloplasty ring.
6. Patients needing emergency or life-saving interventions.
7. Patients with a heavily calcified mitral annulus and/or anterior mitral leaflet.
8. Patients with active infection or endocarditis (suspect endocarditis included).
9. Patients with echocardiographic evidence of intracardiac mass or thrombus.
10. Patients which suffered an acute myocardial infarction within 30 days of the intended treatment (defined as: Q wave MI, or non-Q wave MI with elevation of CK-MB ≥ 3 times normal in the absence of pathological Q waves), if no assay for CK-MB was performed, elevation of CK level to >2 times normal without new Q waves, or elevated Troponin level is also considered a non-Q wave MI).
11. Patients with an active peptic ulcer or upper GI bleeding within the prior 30 days.
12. Patients with a documented allergy towards contrast media, and to any compound of the investigated medical device.
13. Patients that have neurological disease severely affecting ambulation or day to day functioning.
14. Patients with any stroke within the prior 30 days.
15. Patients with senile dementia, according to the advice from a specialized neurologist.
16. Patients in whom transesophageal echocardiography (TEE) is contraindicated since TEE is used for both preoperative screening and guidance during implant procedure.
17. Patients who is unwilling or deemed by the Investigator to be unwilling to comply with the requirements of the protocol, or subject with a history of non-compliance.
18. Patients unable to understand and sign the Informed Consent Form in absence of legal representative.
19. Patients with a lack of capacity to consent.
20. Patients unable to read and write.

    - Echographic exclusion criteria (preoperative screening)
21. Patients with left ventricular apex aneurysm;
22. Patients with aorto-mitral angle <120°;
23. Patients with a systolic/diastolic mitral valve area assessed as not compatible with the sizing policy matrix defined by the Sponsor.

    - Computerized Tomographic (CT) exclusion criteria (preoperative screening)
24. Patients with ventricular morphology (position of papillary muscles, ventricular wall hypertrophy) unsuitable with the study valve design;
25. Patients with aorto-mitral angle <120°;
26. Patients with a systolic/diastolic mitral valve area assessed as not compatible with the sizing policy matrix defined by the Sponsor.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Device Safety | [Timeframe: at 30 days]
  defined as the absence of major device or procedure related serious adverse events evaluated on the following clinical events:
  1. death
  2. major cardiac structural complications (as per MVARC definitions)
  3. life-threatening bleeding (MVARC scale)
  4. any prosthesis-related dysfunction, migration, thrombosis, or other complication, that require surgery or repeated intervention.
  5. myocardial infarction or coronary ischemia requiring PCI or CABG
  6. severe hypotension, heart failure or respiratory failure requiring intravenous vasopressors or invasive or mechanical heart failure treatments such as ultrafiltration or hemodynamic assist devices, including intra-aortic balloon pumps or left ventricular or biventricular assist devices, or prolonged intubation for ≥ 48H
  7. major vascular complications
  8. stroke
  9. stage 2 or 3 acute kidney injury (includes new dialysis)
Device Success | [Timeframe: at 30 days]
  1. Technical Success (as per MVARC definition) defined as alive patient at exit from procedure room, with all of the following:
     1. Successful access, delivery and retrieval of the Epygon delivery system
     2. Successful deployment and positioning of the Epygon Transcatheter mitral valve
     3. Freedom from additional emergency surgery or re-intervention related to the device or access procedure.
  2. Continued intended safety and performance of the device, including:
     1. No evidence of structural or functional failure (as per MVARC definition)
     2. No specific device-related technical failure issues and complications (as per MVARC definition)
     3. Reduction of mitral regurgitation (MR) to either optimal (0+ to trace) or acceptable (reduced by at least 1 grade from baseline with no more than 2+ MR) without significant mitral stenosis (post-procedure EOA ≥ 1.5 cm2 with a transmitral gradient < 5mmHg) and with no greater than mild (1+) paravalvular MR (and without associated hemolysis)

SECONDARY OUTCOMES:
Device Safety | [Time frame: 3, 6, 12 months and yearly up to 5 years from implantation]
  defined as absence of major device or procedure related serious adverse events evaluated on the following clinical events:
  1. death
  2. major cardiac structural complications
  3. life-threatening bleeding (MVARC scale)
  4. any prosthesis-related dysfunction, migration, thrombosis, or other complication, that require surgery or repeated intervention.
  5. myocardial infarction or coronary ischemia requiring PCI or CABG
  6. severe hypotension, heart failure or respiratory failure requiring intravenous vasopressors or invasive or mechanical heart failure treatments such as ultrafiltration or hemodynamic assist devices, including intra-aortic balloon pumps or left ventricular or biventricular assist devices, or prolonged intubation for ≥ 48H
  7. major access complications
  8. stroke
  9. stage 2 or 3 acute kidney injury (includes new dialysis)
Patient success (as per MVARC definition) | [Time frame: 12 months from implantation]
  All of the following must be present:
  1. Device success (either optimal or acceptable)
  2. Patient returned to the pre-procedural setting
  3. No rehospitalizations or reinterventions for the underlying condition (e.g., mitral regurgitation, heart failure)
  4. Improvement from baseline in symptoms (e.g., NYHA improvement by ≥ 1 functional class)
  5. Improvement from baseline in functional status (e.g., 6-min walk test improvement by ≥ 50 m)
  6. Improvement from baseline in quality-of-life (e.g., Kansas City Cardiomyopathy Questionnaire improvement by ≥ 10)
Evaluation of clinical status on the basis of the NYHA functional classification | [Time frame Preoperative, 30 days, 3, 6, 12 months and yearly up to 5 years from implantation]
Six-minute walk test | [Time frame: Preoperative, 30 days, 3, 6, 12 months and yearly up to 5 years from implantation]
Quality of Life score (Kansas City Cardiomyopathy Questionnaire) | [Time frame: Preoperative, 3, 6, 12 months and yearly up to 5 years from implantation]
  The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Hemodynamic performance assessed by echocardiography | [Time frame: Preoperative on native mitral valve, Postoperative, 30 days, 3, 6, 12 months and yearly up to 5 years from implantation]
  1. Prosthetic mean atrio-ventricular ΔP < 5 mm Hg
  2. Prosthetic Effective Orifice Area (EOA) ≥ 1.5 cm2
  3. Mitral valve regurgitation reduction (vs. preoperative) of at least 1 grade and not more than moderate (2+)
  4. Prosthetic paravalvular valve leakage (PVL) not more than mild (1+) without hemolysis
Technical Success (as per MVARC definition) | [Time Frame: immediately after procedure]
  defined as alive patient at exit from procedure room, with all of the following:
  1. Successful access, delivery and retrieval of the Epygon delivery system
  2. Successful deployment and positioning of the Epygon Transcatheter mitral valve
  3. Freedom from additional emergency surgery or re-intervention related to the device or access procedure.
Device Success | [Time frame: 3, 6, 12 months and yearly up to 5 years from implantation]
  1. Technical Success (as per MVARC definition) defined as alive patient at exit from procedure room, with all of the following:
     1. Successful access, delivery and retrieval of the Epygon delivery system
     2. Successful deployment and positioning of the Epygon bioprosthesis
     3. Freedom from additional emergency surgery or re-intervention related to the device or access procedure.
  2. Continued intended safety and performance of the device, including:
     1. No evidence of structural or functional failure (as per MVARC definition)
     2. No specific device-related technical failure issues and complications (as per MVARC definition)
     3. Reduction of mitral regurgitation (MR) to either optimal (0+ to trace) or acceptable (reduced by at least 1 grade from baseline with no more than 2+ MR) without significant mitral stenosis (post-procedure EOA ≥ 1.5 cm2 with a transmitral gradient < 5mmHg) and with no greater than mild (1+) paravalvular MR (and without associated hemolysis)
Procedural Success | [Time frame: 30 days]
  All of the following must be present:
  1. Device success (either optimal or acceptable), And
  2. Absence of major device or procedure related serious adverse events, including:
     1. death
     2. major cardiac structural complications (as per MVARC definitions)
     3. life-threatening bleeding (MVARC scale)
     4. any prosthesis-related dysfunction, migration, thrombosis, or other complication, that require surgery or repeated intervention.
     5. myocardial infarction or coronary ischemia requiring PCI or CABG
     6. severe hypotension, heart failure or respiratory failure requiring intravenous vasopressors or invasive or mechanical heart failure treatments such as ultrafiltration or hemodynamic assist devices, including intra-aortic balloon pumps or left ventricular or biventricular assist devices, or prolonged intubation for ≥ 48H
     7. major vascular complications
     8. stroke
     9. stage 2 or 3 acute kidney injury (includes new dialysis).
Incidence of adverse events | [Time frame: 30 days, 3, 6, 12 months and yearly up to 5 years from implantation]
Incidence of serious adverse events | [Time frame: 30 days, 3, 6, 12 months and yearly up to 5 years from implantation]
Incidence of adverse events related to device | [Time frame: 30 days, 3, 6, 12 months and yearly up to 5 years from implantation]
Incidence of adverse events related to procedure | [Time frame: 30 days, 3, 6, 12 months and yearly up to 5 years from implantation]
Absence of all-cause mortality | [Time frame: 30 days, 3, 6, 12 months and yearly up to 5 years from implantation]

CONTACTS AND LOCATIONS:
Locations (10):
- Austria (2):
  - Medical University of Innsbruck, Innsbruck
  - Medical University of Vienna - Department of Surgery, Division of Cardiac Surgery, Vienna
- Italy (2):
  - Careggi Hospital Florence Italy Largo Brambilla, Florence
  - A.O.U. Citta della Salute e della Scienza di Torino, Torino
- Dedinje Cardiovascular Institute, Belgrade, Serbia
- Spain (5):
  - Hospital German Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen Del Rocio, Seville